CLINICAL TRIAL: NCT04072952
Title: A Phase 1/2, Open Label, Dose Escalation, and Cohort Expansion Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of ARV-471 Alone and in Combination With Palbociclib (IBRANCE®) in Patients With Estrogen Receptor Positive/Human Epidermal Growth Factor Receptor 2 Negative (ER+/HER2-) Locally Advanced or Metastatic Breast Cancer, Who Have Received Prior Hormonal Therapy and Chemotherapy in the Locally Advanced/Metastatic Setting
Brief Title: A Phase 1/2 Trial of ARV-471 Alone and in Combination With Palbociclib (IBRANCE®) in Patients With ER+/HER2- Locally Advanced or Metastatic Breast Cancer
Acronym: mBC
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arvinas Estrogen Receptor, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Arvinas Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARV-471-mBC-101; C4891019 (Other: Pfizer)
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic Breast Cancer; Malignant Neoplasm of the Breast; mBC; ER+/HER2-; Locally Advanced Breast Cancer; ARV-471; Vepdegestrant; Palbociclib; Ibrance
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: Subsequent dose level is determined by the Cohort Review Committee after the initial starting dose cohort and each subsequent dose cohort completes the first 28 days of treatment
  Dose escalation followed by expansion at a Recommended Phase 2 Dose (RP2D) including a combination cohort with palbociclib (IBRANCE®)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARV-471 (Experimental): Parts A and B: ARV-471 administered once daily (QD) or twice daily (BID) for 28 day cycles.
  Interventions: Drug: ARV-471
- ARV-471 and palbociclib (IBRANCE®) (Experimental): Part C: Daily oral dosages of ARV-471 for 28 days in combination with palbociclib (IBRANCE®) for 21 days.
  Interventions: Drug: ARV-471 in combination with palbociclib (IBRANCE®)

INTERVENTIONS:
Drug: ARV-471 — Parts A and B: ARV-471 administered QD or BID for 28 day cycles.
  Arms: ARV-471
Drug: ARV-471 in combination with palbociclib (IBRANCE®) — Part C: Daily oral dosages of ARV-471 for 28 days in combination with palbociclib (IBRANCE®) for 21 days
  Arms: ARV-471 and palbociclib (IBRANCE®)

SUMMARY:
This is a Phase 1/2 dose escalation and cohort expansion study and will assess the safety, tolerability and anti-tumor activity of ARV-471 alone and in combination with palbociclib (IBRANCE®) in patients with estrogen receptor positive/human epidermal growth factor receptor 2 negative (ER+/HER2-) locally advanced or metastatic breast cancer, who have received prior hormonal therapy and chemotherapy in the locally advanced/metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

Part A, Part B, and Part C:

* Patients at least 18 years of age at the time of signing the informed consent.
* Patients must have histologically or cytologically confirmed ER+ and HER2- advanced breast cancer for which standard curative therapy is no longer effective or does not exist.
* Patients must have measurable or non-measurable disease by RECIST criteria (version1.1), with radiologic tumor assessments performed within 28 days of the first dose of therapy.
* Patients must be willing to undergo a core biopsy of accessible tumor within 4 weeks prior to the initiation of study treatment and a follow-up biopsy on treatment for ER immunohistochemistry (IHC) testing and pharmacodynamics (PD) studies. (Patients without accessible tumor tissue may be eligible after discussion with the Medical Monitor.)
* Women must be postmenopausal due to surgical or natural menopause.

Part A:

- Patients must have received at least 2 prior endocrine regimens in any setting (neoadjuvant, adjuvant or advanced/metastatic) a CDK4/6 inhibitor and up to 3 prior regimens of cytotoxic chemotherapy in the locally advanced or metastatic setting.

Part B:

* Patients must have received at least 1 prior endocrine regimen for a minimum of 6 months in the locally advanced or metastatic setting; if more than 1 prior endocrine regimen has been administered, only one of the regimens must have been administered for a minimum of 6 months in the locally advanced or metastatic setting
* Patients must have received a CDK4/6 inhibitor
* Patients must have received up to 1 prior regimen of cytotoxic chemotherapy in the locally advanced or metastatic setting
* Women must be postmenopausal due to surgical or natural menopause.

Part C:

* Patients must have received at least one prior endocrine regimen.
* Patients must have received no more than two prior chemotherapy regimens for advanced disease.
* Women must be postmenopausal due to surgical or natural menopause.

Exclusion Criteria:

Part A, Part B, and Part C:

* Patients with known symptomatic brain metastases requiring steroids (above physiologic replacement doses). Patients with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to first dose of study drug, have discontinued high-dose corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable as judged by the Investigator.
* Receipt of prior anti-cancer or other investigational therapy within 14 days prior to the first administration of study drug.
* Radiation therapy within 4 weeks of first dose of study drug or prior irradiation to >25% of the bone marrow. Palliative radiation for the alleviation of pain due to bone metastasis will be allowed during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of Dose Limiting Toxicities of ARV-471 | 28 Days
  First Cycle Dose limiting toxicities characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug
Part A: Number of Patients with Adverse Events as a measure of safety and tolerability of ARV-471 | First study drug dose through a minimum of 30 calendar Days After Last study drug administration
  Adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug.
Part A: Incidence of laboratory abnormalities as a measure of safety and tolerability of ARV-471 | First study drug dose through a minimum of 30 calendar Days After Last study drug administration
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Part B: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Clinical benefit response rate based on the summation of CRs, PRs and stable disease of 24 weeks duration or longer
Part C: Incidence of Dose Limiting Toxicities of combination ARV-471 + palbociclib | 28 Days
  First cycle dose-limiting toxicities and determination of a maximum tolerated dose (MTD) if applicable among the doses evaluated
Part C: Number of Patients with Adverse Events as a measure of safety and tolerability of combination ARV-471 + palbociclib | First study drug dose through a minimum of 30 calendar Days After Last study drug administration
  Adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug combination
Part C: Incidence of laboratory abnormalities as a measure of safety and tolerability of combination ARV-471 + palbociclib | First study drug dose through a minimum of 30 calendar Days After Last study drug administration
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing

SECONDARY OUTCOMES:
Part A: Assessment of pharmacokinetic (PK) parameter area under the concentration-time curve (AUC). | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of ARV-471
  Concentration-time curve (AUC) for single and multiple dose of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses.
Part A: Assessment of pharmacokinetic parameter maximum concentration (Cmax). | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of ARV-471
  Maximum concentration (Cmax) for single and multiple dose of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses.
Part A: Assessment of pharmacokinetic parameter minimum concentration (Cmin). | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of ARV-471
  Minimum concentration (Cmin) for single and multiple dose of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses.
Part A: Assessment of pharmacokinetic parameter time to maximum concentration (Tmax). | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of ARV-471
  Time to maximum concentration (Tmax) for single and multiple dose of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses.
Part A: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating overall response rate per RECIST 1.1.
Part A: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating clinical benefit response (CBR) rate based on the summation of complete responses (CRs), partial responses (PRs) and stable disease of 24 weeks duration or longer.
Part A: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating disease control rate (complete response, partial response, stable disease).
Part A: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating progression free survival.
Part A: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating duration of response.
Part B: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating overall response rate per RECIST 1.1 in patients with measurable disease at baseline.
Part B: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating duration of response.
Part B: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating progression-free survival.
Part B: Assessment of anti-tumor activity of ARV-471 | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 will be assessed by evaluating overall survival.
Part B: Evaluation of Plasma Concentrations of ARV-471 | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of investigational products]
  To characterize the pre-dose concentrations of ARV-471.
Part B: Evaluation of Safety and Tolerability | First study drug dose through a minimum of 30 calendar Days After Last study drug administration
  Further evaluation of safety and tolerability of ARV-471 will be based on adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug.
Part B: Evaluation of Safety and Tolerability | First study drug dose through a minimum of 30 calendar Days After Last study drug administration
  Further evaluation of safety and tolerability of ARV-471 will be based on Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Part C:Assessment of pharmacokinetic parameter area under the concentration-time curve (AUC) | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of investigational products
  Concentration-time curve (AUC) for single and multiple doses of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses, and of palbociclib when given alone and in combination with ARV-471.
Part C: Assessment of pharmacokinetic parameter maximum concentration (Cmax). | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of investigational products
  Maximum concentration (Cmax) for single and multiple doses of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses, and of palbociclib when given alone and in combination with ARV-471
Part C: Assessment of pharmacokinetic parameter minimum concentration (Cmin). | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of investigational products
  Minimum concentration (Cmin) for single and multiple dose of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses.
Part C: Assessment of pharmacokinetic parameter time to maximum concentration (Tmax) | At predefined intervals throughout the ARV-471 treatment period, up to approximately 4 weeks after last dose of investigational products
  Time to maximum concentration (Tmax) for single and multiple dose of ARV-471 PK parameters will be assessed when applicable after a single dose and after multiple doses.
Part C: Assessment of anti-tumor activity of ARV-471 in combination with palbociclib | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 in combination with palbociclib will be assessed by evaluating overall response rate per RECIST 1.1 in patients with measurable disease at baseline.
Part C: Assessment of anti-tumor activity of ARV-471 in combination with palbociclib | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 in combination with palbociclib will be assessed by evaluating clinical benefit response (CBR) rate based on the summation of complete responses (CRs), partial responses (PRs) and stable disease of 24 weeks duration or longer.
Part C: Assessment of anti-tumor activity of ARV-471 in combination with palbociclib | through study completion, up to approximately 2 years
  Anti-tumor activity of ARV-471 in combination with palbociclib will be assessed by evaluating time to event endpoints: progression free survival, duration of response.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Clinical Trial Site, Palo Alto, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Santa Monica, California
  - Clinical Trial Site, Norwalk, Connecticut
  - Clinical Trial Site, Fort Myers, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, East Brunswick, New Jersey
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No